CLINICAL TRIAL: NCT00734253
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Phase 2b Study to Evaluate the Safety and Efficacy of Pyridorin (Pyridoxamine Dihydrochloride) in Patients With Nephropathy Due to Type 2 Diabetes
Brief Title: Safety and Efficacy Study of Pyridorin in Patients With Nephropathy Due to Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NephroGenex, Inc. (Industry)
Collaborators: Collaborative Study Group (CSG) (Network); Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PYR-210
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2014-05

CONDITIONS: Diabetic Nephropathy
Keywords: Nephropathy; Kidney Disease; Diabetes; Pyridoxamine; Pyridorin; NephroGenex; PYR-210
MeSH Terms: conditions — Diabetic Nephropathies; Kidney Diseases; Diabetes Mellitus | interventions — pyridoxamine dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Pyridorin 150 mg bid
  Interventions: Drug: Pyridoxamine Dihydrochloride
- 2 (Experimental): Pyridorin 300 mg bid
  Interventions: Drug: Pyridoxamine Dihydrochloride
- 3 (Placebo Comparator): Placebo bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridoxamine Dihydrochloride — 150 mg capsules taken orally twice a day for 1-year.
  Arms: 1
Drug: Pyridoxamine Dihydrochloride — 300 mg capsules taken twice a day for 1-year.
  Arms: 2
Drug: Placebo — Placebo capsules taken twice a day for 1-year
  Arms: 3

SUMMARY:
The primary objective of this study is to evaluate the efficacy of two different doses of Pyridorin (150 mg and 300 mg)compared to placebo in retarding the progression of diabetic nephropathy. This will be assessed by measuring the change in serum creatinine and other biomarkers of kidney disease during the course of the 1-year study.

DETAILED DESCRIPTION:
Diabetic kidney disease afflicts about 20% of all diabetics and is the major cause of end-stage renal disease (ESRD). There are an estimated 1.2 million diabetic overt nephropathy patients in the US, and approximately 5.1 million diabetic patients exhibiting signs of developing kidney disease.

Hyperglycemia-induced microvascular disease is the fundamental cause of diabetic kidney disease. More specifically, hyperglycemia perturbs metabolic pathways, particularly in tissues that do not regulate intracellular glucose levels. This favors a broad range of pathogenic oxidative chemistries including the formation of advanced glycation end-products (AGEs), toxic carbonyls, and reactive oxygen species (ROS) that are considered to be the principal causative factors in the development of diabetic microvascular disease.

Pyridorin™ has been shown to inhibit AGE formation and to scavenge ROS and toxic carbonyl compounds in extensive in vitro studies. The therapeutic potential of Pyridorin™ has been demonstrated in vivo by extensive preclinical studies that have been carried out in a number of independent laboratories by prominent investigators. In addition, Pyridorin™ has demonstrated a significant treatment effect in slowing the progression of diabetic nephropathy in two Phase 2 clinical trials. Thus, a solid scientific rationale and clinical evidence exists for the application of Pyridorin™ therapy to slow the progression of diabetic kidney disease.

NephroGenex is initiating a new Phase 2b clinical trial (PYR-210) that is evaluating the safety and efficacy of Pyridorin™ in slowing the progression of overt nephropathy in patients with type 2 diabetes. This trial incorporates the latest discussion with the FDA regarding the use of an approvable surrogate marker that would be subsequently confirmed with hard clinical endpoints.

In this double-blind, placebo-controlled study, eligible type 2 diabetic patients with overt nephropathy will be treated for one year with bid doses of either Pyridorin™ 150 mg, Pyridorin™ 300 mg, or placebo. The primary endpoint in the study is the change in serum creatinine (SCr) from baseline after 1 year of therapy. Secondary 1-year endpoints include the slope of SCr, the change in protein/creatinine ratio (PCR) derived from 24-hour urine collections, and the change from baseline and slope of serum cystatin C.

The patient population studied will be type 2 diabetics with overt nephropathy defined as having a SCr between 1.3 and 3.3 mg/dl in females and between 1.5 and 3.5 mg/dl in males, accompanied by proteinuria in the macroalbuminuric range (PCR at least 1200 mg/g). In order to reduce confounding variables, careful control of blood pressure (BP) will be required. If not yet controlled, each patient's BP will brought to a level that the investigator believes is appropriate for the patient prior to randomization, and this will remain the target BP for that patient for the remainder of the study. Also, patients will be permitted to be on only one ACE inhibitor or angiotensin receptor blocker (ARB) and no other drugs that inhibit the renin-angiotensin-aldosterone axis throughout the study. A run-in period will be required in some patients to achieve the BP and ACEi/ARB requirements.

This study will be conducted with the leadership of the Collaborative Study Group.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients who have given voluntary written consent to participate in this study prior to conducting Screening Visit procedures;
2. Male and female patients 25 years of age or older with a diagnosis of type 2 diabetes; • If a woman is of childbearing potential (WOCBP) she must agree to use appropriate birth control (double barrier methods, hormonal contraceptives, or intrauterine device)for the duration of the study (WOCBP is defined as all women who are not surgically sterile or are not at least 1 year post-menopausal). All WOCBP must have a negative serum pregnancy test at the Screening Visit;
3. At the Screening Visit, ALL patients must have a history of overt diabetic nephropathy, as defined by the following:

   * A SCr measurement of 1.3 mg/dL to 3.3 mg/dL (women) or 1.5 mg/dL to 3.5 mg/dL (men) inclusive, and
   * A 24-hour urine collection PCR ≥1200 mg/g;
4. Patients must be receiving an ACE-I or an ARB, for at least 3 months prior to the Qualifying Visit (Screening Visit for those patients not entering into the Optional Run-in Period), where the dose of the ACE-I or the ARB is considered appropriate for that patient and has been stable for at least 2 months;
5. Patients must be on stable blood pressure medications for 2 months prior to the Qualifying Visit (Screening Visit for those patients not entering into the Optional Run-in Period), with a seated blood pressure at the Qualifying Visit of ≤160/90 mmHg;
6. At the Qualifying Visit (only applies to those patients who enter into the Optional Run-in Period), the following eligibility parameters must be met in order to be randomized:

   * A SCr measurement within 25% of the SCr measurement at the Screening Visit; and
   * A 24-hour urine collection PCR ≥600 mg/g.

EXCLUSION CRITERIA:

1. Patients with type 1 diabetes;
2. Patients with a diagnosis of chronic renal disease other than diabetic renal disease with or without hypertensive renal disease;
3. Patients receiving a renin inhibitor or an aldosterone antagonist or a combination of an ACE-I and an ARB within 2 months of the Qualifying Visit (Screening Visit for those patients not entering into the Optional Run-in Period);
4. Patients with a history of solid organ transplantation;
5. Patients with a history of myocardial infarction, coronary re-vascularization procedures (including percutaneous transluminal coronary angioplasty), cerebrovascular accident ortransient ischemic attack within 1 month prior to the Screening Visit;
6. Patients with a diagnosis of Class III or IV congestive heart failure at any time (as defined by the New York Heart Association);
7. Patients with a history of neoplastic disease (except basal or squamous cell carcinoma of the skin) within 5 years prior to the Screening Visit;
8. Patients with any history of dialysis within 2 years prior to the Screening Visit;
9. Patients in whom dialysis or renal transplantation is anticipated by their physician within 1 year after the Screening Visit;
10. Patients who used SCr altering drugs within 1 month prior to the Screening Visit;
11. Patients who require systemic immunosuppression therapy for >2 weeks (except for inhalant steroids);
12. Patients with clinically significant liver disease or transaminase (alanine aminotransferase and aspartate aminotransferase) levels >2.5 x upper limit of normal measured at the Screening Visit;
13. Patients with bilirubin levels >1.5 x upper limit of normal measured at the Screening Visit;
14. Patients with a history of allergic or other adverse response to vitamin B preparations;
15. Patients who require >50 mg of vitamin B6 daily;
16. Patients who have a history of dysphasia and swallowing disorders;
17. Patients with a history of hypersensitivity to Pyridorin or any of the excipients in the Pyridorin formulation;
18. Patients who have taken pyridoxamine or any other investigational drug within 30 days prior to the Screening Visit, or have participated in a previous Pyridorin trial or another clinical trial within 30 days prior to the Screening Visit;
19. Patients with a current history of drug or alcohol abuse;
20. Patients unlikely to comply with the study protocol (e.g., an inability and unwillingness to participate in adequate training, an uncooperative attitude, inability to return for follow-up visits, or unlikelihood of completing the study);
21. Women who are lactating, pregnant or intend to become pregnant during the course of the study; and
22. Patients who are employees of NephroGenex or its representatives.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in serum creatinine from baseline to end of study. | 1 year

SECONDARY OUTCOMES:
SCr slope, change in PCR, Cystatin C slope and change from baseline. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Edmund J. Lewis, MD, Study Chair — Collaborative Study Group
Locations (1):
- The Collaborative Study Group, Chicago, Illinois, United States